CLINICAL TRIAL: NCT04543123
Title: Effect of Self-administered Transcranial Direct Stimulation in Patients With Major Depressive Disorder: A Prospective, Randomized, Single-blinded Clinical Trial
Brief Title: Effect of Self-administered tDCS in Patients With MDD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jeong-Ho Chae (Other)
Collaborators: Ybrain Inc. (Industry)
Responsible Party: Sponsor-Investigator, Jeong-Ho Chae, Professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: tDCS in MDD
Record Dates: First submitted 2020-08-28; First posted 2020-09-09 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sham tDCS treatment group (Sham Comparator): the current rose slowly for 30 seconds, descended for 30 seconds, and then remained at zero for 29 minutes
  Interventions: Device: tDCS treatment; Drug: Antidepressant Drug(escitalopram)
- active tDCS treatment group (Experimental): 2mA of current was delivered during the 30 minutes of treatment
  Interventions: Device: tDCS treatment; Drug: Antidepressant Drug(escitalopram)

INTERVENTIONS:
Device: tDCS treatment — Participants visited the hospital four times (biweekly for two weeks). During their second visit, a research nurse instructed each participant on use of home-based tDCS equipment (YDS-301N; Ybrain Inc., Seongnam-si, Korea) and all participants thereafter conducted tDCS treatment at home once a day for 30 minutes (five times per week).
Drug: Antidepressant Drug(escitalopram) — Participants in both active and sham groups were prescribed escitalopram in combination with tDCS treatment.

SUMMARY:
In this randomized, single-blinded clinical trial, 58 patients with major depressive disorder were assigned to active and sham tDCS stimulation groups in a 1:1 ratio, and treatment responses were evaluated biweekly over six weeks.

DETAILED DESCRIPTION:
Patients were randomized to receive either real or sham-tDCS as well as anti-depressant drugs. tDCS was applied over the left (anode) and right (cathode) dorsolateral prefrontal cortex (DLPFC). Patients visited the hospital to get tDCS administrations 5 days a week for 2 weeks. They were evaluated every 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of a major depressive disorder as confirmed by the SCID-IV and MINI (without psychotic features)
* Greater than 22 points of Montgomery-Asberg Depression Rating Scale
* Aged 19 to 65.
* Has provided informed consent
* Has received Escitalopram as a combined antidepressant during the study period

Exclusion Criteria:

* Has other mental disorders diagnosed by Axis-I, except major depressive disorder (However, subject who is diagnosed as both major depressive disorder as well as anxiety disorder can participate the study.)
* History of suicidal attempt in the last 6 months
* Diagnosed with bipolar or psychotic major depressive disorder
* Diagnosed with other depressive disorders: dysthymic disorder, and depressive disorders that are not elsewhere classified.
* Has hypersensitivity to Escitalopram ingredients
* A score of 5 or greater for the question #10 in MADRS
* Diagnosed with closed angle glaucoma or has a history of glaucoma.
* History of participation in other clinical trials within 30days.
* A major and/or unstable medical or neurologic illness
* Currently taking substances pimozide
* Pregnant or has a positive pregnancy serum test.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2019-05-02 (Actual); Study Completion 2019-05-02 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Scale (HAM-D) | Change from Baseline Hamilton Depression Scale at 6 weeks
  Hamilton Depression Scale was deployed by a trained psychiatrist at every visit.With a total of 17 questions, the overall score is rated from 0 to 34, and higher total scores indicate more severe depression symptoms

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI) | Weeks 0, 2, 4, and 6
  The self-rated scale of the Beck Depression Inventory (BDI) was completed by participants. With a total of 21 questions, the score is rated from 0 to 33, and higher total scores indicate more severe depression symptoms.
Montgomery-Asberg Depression Rating Scale | Weeks 0, 2, 4, and 6
  Montgomery-Asberg Depression Rating Scale was deployed by a trained psychiatrist at every visit. Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60.
Beck Anxiety Inventory | Weeks 0, 2, 4, and 6
  Beck Anxiety Inventory was deployed by a trained psychiatrist at every visit. The BAI contains 21 questions, each answer being scored on a scale value of 0 (not at all) to 3 (severely). Higher total scores indicate more severe anxiety symptoms. The overall score ranges from 0 to 63.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul St. Mary's Hospital, The Catholic University of Korea, Seoul, South Korea